CLINICAL TRIAL: NCT04956133
Title: Effectiveness and Implementation of Physical Activity for Children and Adolescents on Treatment for Cancer and/or Blood Diseases
Brief Title: IMPACT: IMplementation of Physical Activity for Children and Adolescents on Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other); Stollery Children's Hospital (Other); Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0364
Record Dates: First submitted 2021-06-11; First posted 2021-07-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Cancer; Pediatric Hematology
Keywords: Childhood cancer; Adolescent cancer; In-patient; Out-patient; Oncology; Hematology
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical activity (Experimental): Participants will be offered online, individualized physical activity sessions 2-3 times/week for 15-45 minutes/session for 8-12 weeks.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Participants will receive the IMPACT program, which includes a combination of aerobic, resistance, balance, and flexibility exercises conducted 1:1 and delivered online by a physical activity specialist via Zoom. The IMPACT program follows basic physical activity progression principles (i.e., principles of frequency, intensity, time, type, overload and progression). Tailoring will be used to promote fitness and wellness benefits, while ensuring safety. In addition, prominent behaviour change techniques will be provided by physical activity specialists within each 1:1 session. Discussions and worksheets will be provided, depending on participants needs.

SUMMARY:
Physical activity can enhance well-being among youth diagnosed with oncological or hematological diseases. We developed a tailored, 1:1, online physical activity program (i.e., IMPACT), to promote physical activity in this cohort. The proposed single-group, mixed-methods project will assess the effect of IMPACT and explore markers of implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Children or adolescents between the ages of 5-18 years at enrollment and at least one parent (defined as a caregiver; biological or otherwise)
2. Diagnosed with any oncological and/or hematological diagnosis
3. Currently receiving or scheduled to receive any treatment for any oncological and/or hematological diagnosis or completed treatment <3 months

Exclusion Criteria:

1. Completed all treatment for their oncological or hematological diagnosis >3 months
2. Unable to participate in physical activity as assessed by the patients' healthcare team or physical activity specialist
3. Parent and/or patient cannot understand verbal English
4. Parent is unwilling to be present (i.e., at home, in the same room depending on participant age and functional ability) during the physical activity sessions (required to ensure safety of the child/adolescent)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Reach | Through study completion, an average of 6 years.
  The number of people who participate, and reasons why or why not.

SECONDARY OUTCOMES:
Attendance | Through study completion, an average of 6 years.
  Number of sessions attended out of the number of sessions offered by study staff.
Adherence | Through study completion, an average of 6 years.
  Number of assessments completed out of number of scheduled assessments.
Self-Reported Physical Activity Behaviour | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Modified Leisure Time Exercise Questionnaire (Godin & Shephard, 1985). Time spent in mild, moderate, and vigorous activity will be calculated. Higher numbers indicate greater physical activity.
Directly Assessed Physical Activity Behaviour | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  7-day wear period (minimum) with an activity monitor. Higher numbers indicate greater time spent in physical activity and intensity.
Functional Mobility | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  The timed up and go test (shorter time indicates better functional mobility). Note, this and other "physical tests" to follow were selected based on use with healthy children, children with chronic conditions, and adults with and without chronic conditions (e.g., Bohannon, 1995; Canadian Society of Exercise Physiology, 2019; Deforche et al., 2003; Haas et al., 2017; Jankowski et al., 2015; Kolber & Hanney, 2012; Lemmink et al., 2003; McNeely et al., 2019; Muir et al., 2010; Podsiadlo & Richardson, 1991; Thorsteinsson et al., 2013).
Lower Extremity Endurance | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  30-second sit to stand test (more sit/stands indicates greater lower extremity endurance).
Balance | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Flamingo balance test (longer time without falling, reaching, shuffling/jumping indicates better balance).
Range of Motion | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Shoulder range of motion (ROM; greater number indicates greater ROM).
Flexibility | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  sit and reach flexibility (greater distance indicates higher flexibility).
Aerobic Capacity | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Aerobic step tests (more steps indicates higher aerobic capacity).
Cancer-Specific Quality of Life | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  PedsQL 3.0 Cancer Module (Varni et al., 2009). Score range 0-100; higher scores indicate better quality of life.
Health-Related Quality of Life | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  PedsQL 4.0 Generic Core Scales (Varni et al., 2009). Score range 0-100; higher scores indicate better quality of life.
Symptoms | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Symptom Screening in Pediatrics Tool (Hyslop et al., 2018). Score range 0-60; higher score indicates more symptoms experienced and greater severity of symptoms experienced.
Cognitive Functioning | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Behavior Rating Inventory of Executive Function 2nd Ed (Gioia et al., 2015). Frequency of behaviors are ranked from "Never" to "Often," and results are reported as t scores where higher scores indicate greater deficits.
Maintenance of Physical Activity | Baseline (week 0), post-intervention (week 8-12), 6-month follow-up (week 20-24), 1 year follow-up (week 48-52)
  Number of participants who maintain physical activity following the program.
Physical Activity Fidelity | Through study completion, an average of 6 years.
  Fidelity of the physical activity program implementation will be assessed via randomly video-auditing a subset of sessions.
Time to Implement and Deliver | Through study completion, an average of 6 years.
  Time and expertise to deliver the intervention and physical assessments will be tracked.
Adverse Events | Through study completion, an average of 6 years.
  Adverse events will be defined as any negative effect caused (or suspected to be caused by) the physical activity program.
Healthcare Provider and Staff Uptake | Through study completion, an average of 6 years.
  Healthcare providers' and clinical staffs' referral to the physical activity program

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Thorsteinsson T, Helms AS, Adamsen L, Andersen LB, Andersen KV, Christensen KB, Hasle H, Heilmann C, Hejgaard N, Johansen C, Madsen M, Madsen SA, Simovska V, Strange B, Thing LF, Wehner PS, Schmiegelow K, Larsen HB. Study protocol: Rehabilitation including Social and Physical activity and Education in Children and Teenagers with Cancer (RESPECT). BMC Cancer. 2013 Nov 14;13:544. doi: 10.1186/1471-2407-13-544. PMID 24229362
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Deforche B, Lefevre J, De Bourdeaudhuij I, Hills AP, Duquet W, Bouckaert J. Physical fitness and physical activity in obese and nonobese Flemish youth. Obes Res. 2003 Mar;11(3):434-41. doi: 10.1038/oby.2003.59. PMID 12634442
- [Background] Canadian Society of Exercise Physiology. (2019). The CSEP physical activity training for health resource manual, 2nd edition.
- [Background] McNeely ML, Sellar C, Williamson T, Shea-Budgell M, Joy AA, Lau HY, Easaw JC, Murtha AD, Vallance J, Courneya K, Mackey JR, Parliament M, Culos-Reed N. Community-based exercise for health promotion and secondary cancer prevention in Canada: protocol for a hybrid effectiveness-implementation study. BMJ Open. 2019 Sep 13;9(9):e029975. doi: 10.1136/bmjopen-2019-029975. PMID 31519676
- [Background] Muir SW, Corea CL, Beaupre L. Evaluating change in clinical status: reliability and measures of agreement for the assessment of glenohumeral range of motion. N Am J Sports Phys Ther. 2010 Sep;5(3):98-110. PMID 21589666
- [Background] Lemmink KA, Kemper HC, de Greef MH, Rispens P, Stevens M. The validity of the sit-and-reach test and the modified sit-and-reach test in middle-aged to older men and women. Res Q Exerc Sport. 2003 Sep;74(3):331-6. doi: 10.1080/02701367.2003.10609099. No abstract available. PMID 14510299
- [Background] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645
- [Background] Jankowski M, Niedzielska A, Brzezinski M, Drabik J. Cardiorespiratory fitness in children: a simple screening test for population studies. Pediatr Cardiol. 2015 Jan;36(1):27-32. doi: 10.1007/s00246-014-0960-0. Epub 2014 Jul 29. PMID 25070386
- [Background] Haas F, Sweeney G, Pierre A, Plusch T, Whiteson J. Validation of a 2 minute step test for assessing functional improvement. Open J Therap Rehab. 2017;5(02):71.
- [Background] Varni JW, Limbers CA. The pediatric quality of life inventory: measuring pediatric health-related quality of life from the perspective of children and their parents. Pediatr Clin North Am. 2009 Aug;56(4):843-63. doi: 10.1016/j.pcl.2009.05.016. PMID 19660631
- [Background] Hyslop S, Dupuis LL, Baggott C, Dix D, Gibson P, Kuczynski S, Johnston DL, Orsey A, Portwine C, Price V, Spiegler B, Tomlinson D, Vanan M, Tomlinson GA, Sung L. Validation of the Proxy Version of Symptom Screening in Pediatrics Tool in Children Receiving Cancer Treatments. J Pain Symptom Manage. 2018 Jul;56(1):107-112. doi: 10.1016/j.jpainsymman.2018.03.025. Epub 2018 Apr 6. PMID 29630923
- [Background] Gioia GA, Issquith PK, Guy SC, Kenworthy L. Behavior Rating Inventory of Executive Function®, Second Edition (BRIEF®2). 2015. Lutz, FL: PAR Inc.
- [Derived] McLaughlin E, Culos-Reed SN, Chamorro-Vina C, Wilson B, Fisher S, Guilcher GM, Penney B, Penney M, Wich L, Wich J, Wurz A. IMplementation of Physical Activity for Children and adolescents on Treatment (IMPACT) for Cancer Diagnoses in Alberta: Protocol for a Single-Arm, Mixed-Methods, Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2025 Dec 17;14:e59302. doi: 10.2196/59302. PMID 41406465